CLINICAL TRIAL: NCT01733316
Title: A Long-Term, Open-Label, Safety, Tolerability and Superior Effectiveness Study of Cysteamine Bitartrate Delayed-release Capsules (RP103) in Patients With Cystinosis
Brief Title: Open-Label, Safety and Superior Effectiveness Study of Cysteamine Bitartrate Delayed-Release Capsules (RP103) in Cystinosis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RP103-07; 2012-002773-64 (EudraCT Number)
Record Dates: First submitted 2012-11-16; First posted 2012-11-27 (Estimated); Results first posted 2017-05-24 (Actual); Last update posted 2024-12-27 (Actual); Status verified 2024-12

CONDITIONS: Cystinosis
Keywords: Nephropathic Cystinosis; Cysteamine; Delayed-Release Cysteamine; Orphan Disease; CTNS Protein, Human
MeSH Terms: conditions — Cystinosis; Rare Diseases | interventions — Cysteamine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- All Participants (Experimental): Cystagon® Phase: From Screening and during Months 1, 2, 3 participants receive their usual dose of Cystagon® every 6 hours (Q6H).
  RP103 Phase: During Months 3.5, 4, 5, 6, 7 participants receive RP103 every 12 hours (Q12H).
  Long Term Phase: On or after Month 7, for the remainder of study participants receive RP103 Q12H.
  Interventions: Drug: RP103; Drug: Cystagon®

INTERVENTIONS:
Drug: RP103
  Other Names: cysteamine bitartrate delayed-release capsules; PROCYSBI®
Drug: Cystagon®
  Other Names: cysteamine bitartrate

SUMMARY:
The purpose of this study is to gather information about the effectiveness (how well it works to treat cystinosis) and safety of a new form of cysteamine bitartrate called RP103, compared to the already-approved drug cystinosis patients are taking called Cystagon®.

In cystinosis, the body builds up cystine. When taken regularly, the active ingredient of Cystagon® (cysteamine bitartrate) reduces cystine in the body. RP103 has the same active ingredient as Cystagon® and is designed to reduce cystine in a similar way that Cystagon® does. To decide if RP103 is better than Cystagon®, the study will look at two types of blood tests. One test is pharmacodynamics (PD), which measures the amount of white blood cell (WBC) cystine after taking study drug. WBC cystine is a laboratory test used to find out if cysteamine bitartrate is reducing cystine levels in the body. The second test is pharmacokinetics (PK), which measures the amount of cysteamine in the blood after taking the drug.

RP103 is different from Cystagon®: Instead of the cysteamine bitartrate being absorbed from the stomach, RP103 is designed to be absorbed from the small intestine. This may make the effects of the drug last longer, so that it can be taken twice a day instead of four times a day like Cystagon®.

Some cystinosis patients have bad breath (halitosis) when they take Cystagon®. Study participants who experience bad breath with Cystagon® will be asked if they would like to participate in an optional "halitosis substudy" to investigate this issue by collecting some extra PK blood samples.

DETAILED DESCRIPTION:
Study with completed results acquired from Horizon in 2024.

ELIGIBILITY:
INCLUSION CRITERIA:

* Male or female with a documented diagnosis of cystinosis
* On a stable dose of Cystagon® at least 21 days prior to Screening
* WBC cystine level > 1 nmol 1/2 cystine/mg of protein, on average over at least 2 measurements collected during the 2 years prior to Screening
* No clinically significant change in liver function tests, i.e. 1.5 times upper limit of normal (ULN) for alanine aminotransferase and aspartate aminotransferase, and/or 1.5 times ULN for total bilirubin, within 6 months prior to Screening
* No clinically significant change in renal function, i.e. estimated glomerular filtration rate (GFR) within 6 months prior to Screening
* Must have an estimated GFR > 20 mL/minute/1.73m^2 (using the equation from Schwartz 2009 J Am Soc Nephrol 20:629-647)
* Female subjects who are sexually active and of childbearing potential, i.e. not surgically sterile (tubal ligation, bilateral oophorectomy, or hysterectomy) or at least 2 years naturally postmenopausal must agree to use an acceptable form of contraception from Screening through completion of the study. Acceptable forms of contraception for this study include hormonal contraceptives (oral, implant, transdermal patch, or injection) at a stable dose for at least 3 months prior to Screening, barrier (spermicidal condom or diaphragm with spermicide), intrauterine device, or a partner who has been vasectomized for at least 6 months.
* Subject or their parent or guardian must provide written informed consent, assent (where applicable), prior to participation in the study

EXCLUSION CRITERIA:

* Younger than 12 years of age
* Current history of the following conditions or any other health issues that make it, in the opinion of the investigator, unsafe for study participation:

  * Inflammatory bowel disease, if currently active, or prior resection of the small intestine;
  * Heart disease (e.g., myocardial infarction, heart failure, unstable arrhythmias, or poorly controlled hypertension) within 90 days prior to Screening;
  * Active bleeding disorder within 90 days prior to Screening;
  * History of malignant disease within 2 years prior to Screening
* Hemoglobin level of < 9 g/dL at Screening or, in the opinion of the investigator, a hemoglobin level that would make it unsafe for study participation
* Known hypersensitivity to cysteamine and penicillamine
* Female subjects who are nursing, planning a pregnancy, or are known or suspected to be pregnant
* Subjects who, in the opinion of the investigator, are not able or willing to comply with study requirements.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2013-01-31 (Actual); Primary Completion 2015-02 (Actual); Study Completion 2017-07-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (14):
- United States (5):
  - California Pacific Medical Center (CPMC) Research Institute, San Francisco, California
  - Stanford University Medical School, Stanford, California
  - Emory Children's Center, Atlanta, Georgia
  - Ann & Robert H. Lurie Children's Hospital of Chicago, Chicago, Illinois
  - Baylor College of Medicine / Texas Childrens Hospital, Houston, Texas
- University Hospital of Leuven, Leuven, Belgium
- France (3):
  - Hospices Civils de Lyon, Lyon
  - Hôpital Necker-Enfants Malades, Paris
  - Hôpital Robert Debré, Paris
- Ospedale Pediatrico Bambino Gesù, Rome, Italy
- Radboud University Nijmegen Medical Center, Nijmegen, Netherlands
- United Kingdom (3):
  - Queen Elizabeth Hospital Birmingham, Birmingham
  - Great Ormond Street, London
  - Guy's Hospital, London

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Schwartz GJ, Munoz A, Schneider MF, Mak RH, Kaskel F, Warady BA, Furth SL. New equations to estimate GFR in children with CKD. J Am Soc Nephrol. 2009 Mar;20(3):629-37. doi: 10.1681/ASN.2008030287. Epub 2009 Jan 21. PMID 19158356
- See also: RP103 (marketed as PROCYSBI) is now approved by the US FDA for management of nephropathic cystinosis in patients 6 years and older. — http://procysbi.com/

RESULTS

PARTICIPANT FLOW:
Groups:
- All Participants: Cystagon® Phase: From Screening and during Months 1, 2, 3 participants received their usual dose of Cystagon® every 6 hours (Q6H).
  RP103 Phase: During Months 3.5, 4, 5, 6, 7 participants received RP103 every 12 hours (Q12H).
  Long Term Phase: On or after Month 7, for the remainder of study participants received RP103 Q12H.
Period: Cystagon® Phase
Arm/Group | All Participants
Started | 41
Completed | 41
Not Completed | 0
Period: RP103 Phase
Arm/Group | All Participants
Started | 41
Completed | 40
Not Completed | 1
Not completed — Non-compliance | 1
Period: Long Term Extension Phase
Arm/Group | All Participants
Started | 38 (Two participants did not enter the long term follow up period.)
Completed | 33
Not Completed | 5
Not completed — Adverse Event | 1
Not completed — Consent Withdrawn by Subject | 2
Not completed — Sponsor Decision | 2

BASELINE CHARACTERISTICS:
Groups:
- All Participants: Cystagon® Phase: From Screening and during Months 1, 2, 3 participants received their usual dose of Cystagon® Q6H.
  RP103 Phase: During Months 3.5, 4, 5, 6, 7 participants received RP103 Q12H.
  Long Term Phase: On or after Month 7, for the remainder of study participants received RP103 Q12H.
Arm/Group | All Participants
Number analyzed (Participants) | 41
Age, Continuous [Mean (Standard Deviation); unit: years] | 24.5 (11.56)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21
  Male | 20

OUTCOME MEASURES:

1. Primary Outcome: Average Difference Between Morning and Non-Morning Log White Blood Cell (WBC) Cystine Values
Description: The primary analysis of WBC cystine was performed using the natural log transformed WBC cystine level; the log transformation is a normalizing transformation. For each participant, the difference between the morning and corresponding non-morning log WBC cystine value (non-morning minus morning) at each monthly visit during the Cystagon® phase (Months 1, 2, and 3) was computed and these differences were averaged. The average difference between morning and non-morning log WBC cystine value was similarly computed for each participant during the RP103 phase (Months 5, 6, and 7). The primary analysis compared within-subject pairs (Cystagon® phase paired with RP103 phase) of non-morning minus morning average differences of log WBC cystine level.
Time Frame: While taking Cystagon® (Months 1, 2, 3): within 15 minutes pre-morning (AM) and pre-non AM dose. During 3 months of RP103 (Months 5, 6, 7): 30 minutes post-AM and post-evening (PM) dose.
Population: Pharmacodynamic (PD) Analysis Set: All participants who received at least one treatment of Cystagon® and RP103 and who had at least one WBC cystine level recorded after each of Cystagon® treatment and RP103 treatment. Only participants with an average difference during both the Cystagon® and RP103 phases were included.
Measure: Mean (Standard Deviation); unit: log [nmol ½ cystine/mg protein]
Groups:
- Cystagon® Phase: From Screening and during Months 1, 2, 3: participants received their usual dose of Cystagon® Q6H.
- RP103 Phase: During Months 3.5, 4, 5, 6, 7: participants received RP103 Q12H.
Arm/Group | Cystagon® Phase | RP103 Phase
Number analyzed (Participants) | 40 | 40
log [nmol ½ cystine/mg protein] | -0.229 (0.5027) | 0.080 (0.3939)
Statistical Analysis 1: Comparison: Cystagon® Phase vs RP103 Phase; Test type: Superiority; p = 0.0048, Paired t-test, two-sided — Paired t-test testing the null hypothesis that the population average difference during the Cystagon® phase is equal to the population average difference during the RP103 phase

2. Secondary Outcome: Number of Participants With Treatment-Emergent Adverse Events (AEs), Serious Adverse Events (SAEs), and Discontinuations Due to AEs
Description: AE: any untoward medical occurrence that does not necessarily have a causal relationship with study drug. SAE: any untoward medical occurrence that at any dose: results in death; is life threatening; requires inpatient hospitalization or prolongation of existing hospitalization; results in persistent or significant disability or incapacity; is a congenital anomaly or birth defect; or is medically significant, and though not included in the above list, is an important medical event, according to the Investigator. Treatment-emergent adverse events (TEAEs) occurred after first dose of study drug. Clinically significant abnormalities in laboratory values (hematology, blood chemistry, urinalysis), electrocardiograms (ECGs), vital signs, and physical examinations were to be reported as adverse events and so are included in this summary of TEAEs
Time Frame: From first dose of study drug to 7 days after last dose. Median duration of exposure was 91 days (range 82-108) for Cystagon® phase, 119 days (range 98-137) for the RP103 phase, and 861 days (range 30 - 1350) during the long-term RP-103 phase.
Population: Safety Analysis Set: all participants who received at least 1 dose of study drug (RP103). The row "At least 1 TEAE" includes both serious and non-serious AEs.
Measure: Count of Participants; unit: Participants
Groups:
- Cystagon® Phase: From Screening and during Months 1, 2, 3: participants received their usual dose of Cystagon® Q6H.
  Observations from Day 1 Cystagon® dosing up to the first dose of RP103 were attributed to the Cystagon® Phase.
- RP103 Phase: During Months 3.5, 4, 5, 6, 7: participants received RP103 Q12H.
  Observations on or after the first dose of RP103 up to Month 7 or study termination visit (whichever occurred first) were attributed to the RP103 Phase.
- Long-Term Phase: From Month 7 and for the remainder of study: participants received RP103 Q12H.
  Observations on or after the Month 7 visit through study termination were attributed to the Long-Term RP103 Phase.
Arm/Group | Cystagon® Phase | RP103 Phase | Long-Term Phase
Number analyzed (Participants) | 41 | 41 | 38
Participants
  At least 1 TEAE | 31 | 38 | 32
  At least 1 TEAE-related to study drug | 4 | 20 | 18
  At least 1 grade ≥ 3 TEAE | 5 | 4 | 13
  At least 1 serious TEAE | 5 | 6 | 13
  At least 1 TEAE leading to discontinuation | 0 | 0 | 1

3. Secondary Outcome: Halitosis Substudy: Maximum Plasma Concentration (Cmax) for Plasma Cysteamine
Description: Participants who reported halitosis ("bad breath") as a side effect while receiving Cystagon® were asked to participate in a substudy to investigate the concentration of dimethylsulfide (DMS) in expired air after the administration of study medication. To assess halitosis during study medication treatment, the steady state pharmacokinetic (PK) samples of cysteamine and DMS were collected over a 6 hour period when Cystagon® was administered and over a 12 hour period when RP103 was administered.
Time Frame: While taking Cystagon® (Month 1, 2 or 3): Within 15 minutes prior to morning dose, 30 minutes post-dose, 1, 2, 4 and 6 hours post-dose. While taking RP103 (Month 5, 6, or 7): 30 minutes after morning dose and 1, 2, 3, 4, 6, 8, 10, 12 hours post-dose
Population: PK Analysis Set: All participants who received at least one dose of RP103 and had available PK data at given timepoint.
Measure: Mean (Standard Deviation); unit: mg/L
Groups:
- Halitosis Substudy Participants: Cystagon® Phase: From Screening and during Months 1, 2, 3 participants received their usual dose of Cystagon® Q6H.
  RP103 Phase: During Months 3.5, 4, 5, 6, 7 participants received RP103 Q12H.
Arm/Group | Halitosis Substudy Participants
Number analyzed (Participants) | 20
mg/L
  Cystagon® dosing period: number analyzed (Participants) | 19
  Cystagon® dosing period | 3.5 (1.87)
  RP103 dosing period | 2.9 (1.65)

4. Secondary Outcome: Halitosis Substudy: Time to Cmax (Tmax) for Plasma Cysteamine
Description: Participants who reported halitosis ("bad breath") as a side effect while receiving Cystagon® were asked to participate in a substudy to investigate the concentration of DMS in expired air after the administration of study medication. To assess halitosis during study medication treatment, the steady state PK samples of cysteamine and DMS were collected over a 6 hour period when Cystagon® was administered and over a 12 hour period when RP103 was administered.
Time Frame: as for outcome 3
Population: PK Analysis Set: All participants who received at least one dose of RP103 and had available PK data at given timepoint.
Measure: Mean (Standard Deviation); unit: hour
Arm/Group | Halitosis Substudy Participants
Number analyzed (Participants) | 20
hour
  Cystagon® dosing period: number analyzed (Participants) | 19
  Cystagon® dosing period | 1.2 (0.87)
  RP103 dosing period | 3.2 (1.30)

5. Secondary Outcome: Area Under the Plasma Concentration Time Curve From Time Point 0 Through the Last Measurable Point (AUC0-t) for Plasma Cysteamine
Description: as for outcome 4
Time Frame: as for outcome 3
Population: PK Analysis Set: All participants who received at least one dose of RP103 and had available PK data at given timepoint.
Measure: Mean (Standard Deviation); unit: hr*mg/L
Arm/Group | Halitosis Substudy Participants
Number analyzed (Participants) | 20
hr*mg/L
  Cystagon® dosing period: number analyzed (Participants) | 19
  Cystagon® dosing period | 7.8 (5.18)
  RP103 dosing period | 9.4 (4.86)

6. Secondary Outcome: Halitosis Substudy: Expired Air DMS Concentrations
Description: as for outcome 4
Time Frame: While taking Cystagon® (Month 1, 2 or 3): Within 15 minutes prior to morning dose 30 min post-dose, 2, 3, 4 and 6 hours post-dose. While taking RP103 (Month 4, 5, or 7): Within 15 min. prior to morning dose. 1, 2, 3, 4, 5, 6, 8, 10, 12 hours post dose
Population: PK Analysis Set: All participants who received at least one dose of RP103 and had available PK data at given timepoint.
Measure: Mean (Standard Deviation); unit: nmol/L
Arm/Group | Halitosis Substudy Participants
Number analyzed (Participants) | 20
nmol/L
  Cystagon®, within 15 minutes prior to dose: number analyzed (Participants) | 18
  Cystagon®, within 15 minutes prior to dose | 4.7 (5.54)
  Cystagon®, 30 minutes post dose: number analyzed (Participants) | 18
  Cystagon®, 30 minutes post dose | 4.7 (4.75)
  Cystagon®, 1 hour post morning dose: number analyzed (Participants) | 18
  Cystagon®, 1 hour post morning dose | 6.9 (6.75)
  Cystagon®, 2 hours post morning dose: number analyzed (Participants) | 18
  Cystagon®, 2 hours post morning dose | 11.9 (11.26)
  Cystagon®, 3 hours post morning dose: number analyzed (Participants) | 18
  Cystagon®, 3 hours post morning dose | 11.2 (13.32)
  Cystagon®, 4 hours post morning dose: number analyzed (Participants) | 18
  Cystagon®, 4 hours post morning dose | 8.8 (12.05)
  Cystagon®, 6 hours post morning dose: number analyzed (Participants) | 18
  Cystagon®, 6 hours post morning dose | 4.4 (3.77)
  RP103, within 15 minutes prior to dose | 4.6 (6.05)
  RP103, 1 hour post morning dose | 5.4 (7.71)
  RP103, 2 hours post morning dose | 5.1 (6.28)
  RP103, 3 hours post morning dose | 7.7 (8.53)
  RP103, 4 hours post morning dose | 8.6 (11.22)
  RP103, 5 hours post morning dose | 11.2 (15.86)
  RP103, 6 hours post morning dose | 8.5 (13.87)
  RP103, 8 hours post morning dose | 5.7 (10.76)
  RP103, 10 hours post morning dose | 5.2 (8.13)
  RP103, 12 hours post morning dose | 4.3 (5.32)

ADVERSE EVENTS:
Time Frame: From first dose of study drug to 7 days after last dose. Median duration of exposure was 91 days (range 82-108) for Cystagon® phase, 119 days (range 98-137) for the RP103 phase, and 861 days (range 30-1350) during the long term RP-103 phase.
Groups:
- Long-Term Phase: From Month 7 and for the remainder of study: participants received RP103 Q12H.
Arm/Group | Cystagon® Phase | RP103 Phase | Long-Term Phase
All-Cause Mortality (participants affected / at risk) | 0/41 | 0/41 | 1/38
Serious Adverse Events (participants affected / at risk) | 5/41 | 6/41 | 13/38
Other Adverse Events (participants affected / at risk) | 28/41 | 33/41 | 32/38
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cystagon® Phase (N=41) | RP103 Phase (N=41) | Long-Term Phase (N=38)
Abdominal pain (Gastrointestinal disorders) | 1 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 1 | 2
Chest pain (General disorders) | 0 | 0 | 1
Death (General disorders) | 0 | 0 | 1
Malaise (General disorders) | 0 | 0 | 2
Bacteraemia (Infections and infestations) | 0 | 1 | 0
Cellulitis (Infections and infestations) | 0 | 0 | 1
Diverticulitis (Infections and infestations) | 1 | 0 | 0
Gastroenteritis (Infections and infestations) | 0 | 1 | 2
Lung infection (Infections and infestations) | 0 | 0 | 1
Pneumonia (Infections and infestations) | 1 | 0 | 1
Sepsis (Infections and infestations) | 1 | 0 | 1
Septic shock (Infections and infestations) | 1 | 0 | 0
Urinary tract infection (Infections and infestations) | 1 | 1 | 0
Arteriovenous fistula operation (Surgical and medical procedures) | 1 | 0 | 0
Depression (Psychiatric disorders) | 0 | 0 | 1
Psychotic disorder (Psychiatric disorders) | 0 | 1 | 0
Arteriovenous fistula thrombosis (Injury, poisoning and procedural complications) | 0 | 0 | 1
Procedural hypotension (Injury, poisoning and procedural complications) | 0 | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 4
Hyperkalemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Scoliosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Migraine with aura (Nervous system disorders) | 0 | 0 | 1
Renal failure acute (Renal and urinary disorders) | 0 | 0 | 1
Testicular pain (Reproductive system and breast disorders) | 0 | 0 | 1
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Hypertension (Vascular disorders) | 0 | 0 | 1
Peripheral artery thrombosis (Vascular disorders) | 0 | 0 | 1
Arteriovenous fistula aneurysm (Injury, poisoning and procedural complications) | 0 | 0 | 1
Ossiculoplasty (Surgical and medical procedures) | 0 | 0 | 1
Renal transplant (Surgical and medical procedures) | 0 | 0 | 2
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Fatigue (General disorders) | 0 | 0 | 1
Pyrexia (General disorders) | 0 | 0 | 1
Arteriovenous fistula site complication (Injury, poisoning and procedural complications) | 0 | 1 | 2
Arteriovenous fistula site haemorrhage (Injury, poisoning and procedural complications) | 0 | 1 | 1
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Cerebral haemorrhage (Nervous system disorders) | 0 | 0 | 1
Dizziness (Nervous system disorders) | 0 | 0 | 1
Headache (Nervous system disorders) | 0 | 0 | 1
Loss of consciousness (Nervous system disorders) | 0 | 0 | 1
Syncope (Nervous system disorders) | 0 | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 0 | 2
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Gastroenteritis norovirus (Infections and infestations) | 0 | 0 | 1
Gastroenteritis viral (Infections and infestations) | 0 | 0 | 1
Graft infection (Infections and infestations) | 0 | 0 | 1
Onychomycosis (Infections and infestations) | 1 | 0 | 0
Tonsillitis (Infections and infestations) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Cystagon® Phase (N=41) | RP103 Phase (N=41) | Long-Term Phase (N=38)
Anaemia (Blood and lymphatic system disorders) | 0 | 1 | 4
Conjunctivitis (Eye disorders) | 0 | 1 | 3
Abdominal pain (Gastrointestinal disorders) | 1 | 3 | 5
Abdominal pain upper (Gastrointestinal disorders) | 2 | 6 | 3
Constipation (Gastrointestinal disorders) | 0 | 2 | 3
Diarrhoea (Gastrointestinal disorders) | 4 | 9 | 7
Nausea (Gastrointestinal disorders) | 4 | 15 | 5
Vomiting (Gastrointestinal disorders) | 2 | 11 | 7
Influenza like illness (General disorders) | 0 | 0 | 4
Malaise (General disorders) | 3 | 1 | 1
Pyrexia (General disorders) | 2 | 2 | 2
Bronchitis (Infections and infestations) | 0 | 1 | 2
Candidiasis (Infections and infestations) | 0 | 1 | 2
Ear infection (Infections and infestations) | 0 | 0 | 3
Gastroenteritis (Infections and infestations) | 1 | 4 | 4
Influenza (Infections and infestations) | 0 | 0 | 4
Nasopharyngitis (Infections and infestations) | 8 | 5 | 6
Respiratory tract infection (Infections and infestations) | 1 | 2 | 2
Upper respiratory tract infection (Infections and infestations) | 3 | 0 | 6
Urinary tract infection (Infections and infestations) | 2 | 3 | 4
Viral infection (Infections and infestations) | 1 | 2 | 2
Viral upper respiratory tract infection (Infections and infestations) | 0 | 0 | 2
Blood creatinine increased (Investigations) | 0 | 1 | 2
Hepatic enzyme increased (Investigations) | 0 | 0 | 2
Weight decreased (Investigations) | 1 | 1 | 3
Dehydration (Metabolism and nutrition disorders) | 1 | 0 | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2
Knee deformity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2
Headache (Nervous system disorders) | 8 | 6 | 7
Renal impairment (Renal and urinary disorders) | 0 | 1 | 2
Dysmenorrhoea (Reproductive system and breast disorders) | 0 | 1 | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 3
Skin lesion (Skin and subcutaneous tissue disorders) | 0 | 0 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Horizon requests that any investigator/institution that plans on presenting/publishing results provide written notification of their request 60 days prior to their presentation/publication. Horizon requests that no presentation/publication will be instituted until 12 months after a study is completed, or after the first presentation/publication whichever occurs first. A delay may be proposed of a presentation/publication if Horizon needs to secure patent or proprietary protection.